CLINICAL TRIAL: NCT06821971
Title: Study of Risk Factors for Therapeutic Failure in Chronic Non-Infectious Uveitis After First-Line Immunosuppressive Therapy
Acronym: FAIL-UVEITIS
Status: Active, not recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2025_843_0012
Record Dates: First submitted 2025-01-28; First posted 2025-02-12 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-01

CONDITIONS: Uveitis
Keywords: Uveitis
MeSH Terms: conditions — Uveitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Uveitis is an inflammatory disease of the uvea, constituting the 4th leading cause of legal blindness worldwide and the 3rd leading cause of avoidable blindness . It is not a rare condition, with an incidence of 17 to 52 per 100,000 population and a prevalence of 38 to 204 per 100,000 population. In the case of cortico-dependence, it is generally accepted to propose sparing with a conventional immunosuppressant, whose efficacy is estimated at around 70%, compared with biotherapies, which are considered more effective (over 90%) but only available as 2nd-line treatment. However, there are few studies on the failure factors of this first-line treatment, such as macular thickness , gender, or vitamin D deficiency. Risk factors for flare-ups are nevertheless known, notably ethnicity, and smoking. The aim of this study is to identify risk factors for treatment failure after three months of first-line immunosuppressive therapy in patients with chronic non-infectious uveitis at Amiens-Picardie University Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Age : > 18 years old
* Uveitis requiring immunosuppressive therapy.
* Including at least one posterior involvement according to the SUN terminology: posterior, or intermediate and posterior, or anterior and posterior, or panuveitis.

Exclusion Criteria:

* Uveitis associated with multiple sclerosis or systemic lupus erythematosus.
* Ocular involvement in Behcet's disease requiring biologic therapy as first-line immunosuppressive treatment.
* Uveitis without posterior segment involvement.
* Infectious uveitis.
* Patients objecting to the use of their personal data for research purposes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retrospective cohort study based on medical records of patients who received first-line immunosuppressive (IS) therapy for their uveitis. Patients with chronic non-infectious uveitis at Amiens-Picardie University Hospital, over the period from January 2013 to January 2023.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-01-14 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Number of therapeutic failure at 4 months | 4 months
  Therapeutic failure at 4 months following the initiation of a first-line immunosuppressant in patients with chronic non-infectious uveitis (CNIU).

SECONDARY OUTCOMES:
Number of therapeutic failure at 9 months | 9 months
  Therapeutic failure at 9 months following the initiation of a first-line immunosuppressant in patients with chronic non-infectious uveitis (CNIU).

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens-Picardie, Salouël, France

IPD SHARING:
Plan to Share IPD: No